CLINICAL TRIAL: NCT00010452
Title: Treatment of Cystic Hygroma (Lymphangiomas) in Children- Picibanil(OK432) Sclerotherapy-Multicenter Trial
Brief Title: Study of Picibanil (OK432) Sclerotherapy in Children With Macrocystic Lymphatic Malformations
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Richard JH Smith, MD, University of Iowa Health Care
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199/15706; UIHC-FDR001774
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2008-01

CONDITIONS: Lymphatic Malformations
Keywords: cystic hygroma; lymphangiomas; lymphatic malformations
MeSH Terms: conditions — Lymphatic Abnormalities; Lymphangioma, Cystic; Lymphangioma | interventions — Picibanil

INTERVENTIONS:
Drug: picibanil — Up to .2 mg per injection, given intralesionally every 6-8 weeks
  Other Names: OK432

SUMMARY:
OBJECTIVES:

I. Determine the efficacy of picibanil sclerotherapy in children with macrocystic lymphangioma.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a multicenter study. Patients are stratified according to prior treatment (no prior treatment vs prior surgical treatment) and geographic area.

Patients who meet all study criteria are put in the "Immediate Treatment Group." Patients receive an intralesional injection of picibanil (OK432) with the aid of ultrasonography or transillumination for localization of cysts. Treatment repeats every 6-8 weeks for a total of up to 4 injections.

After completion of treatment, patients are followed at 6 months, 1 year, and 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of macrocystic lymphangioma of the head and/or neck Cystic spaces at least 2.0 mL confirmed by radiographic imaging (MRI or CT) Mixed lymphangiomas (macrocystic and microcystic disease) allowed if macrocystic component comprises at least 50% of the total disease burden
* No mixed hemangioma-lymphangioma lesions
* At least 6 months since prior surgery for lymphangioma

--Patient Characteristics--

* Hematopoietic: No clinically significant hematologic disease No hemodynamic instability
* Hepatic: No clinically significant hepatic disorder
* Renal: No clinically significant renal disease No personal or family history of post-streptococcal glomerulonephritis
* Cardiovascular: No personal or family history of rheumatic heart disease
* Pulmonary: No respiratory failure

Other:

* Not pregnant or nursing
* Negative pregnancy test
* No history of allergy to penicillin
* No concurrent temperature of 100.5 degrees or greater
* No active upper respiratory infection
* No personal or family history of obsessive-compulsive or tic disorders
* No personal or family history of PANDA (pediatric autoimmune neuro- psychiatric disorder associated with streptococcal infections)
* No history of hypersensitivity to iodine, Omnipaque, or gadolinium (if fluoroscopy is considered necessary)
* No history of poor health (including congenital disorders, chronic diseases, or immunologic dysfunction)

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2000-04; Primary Completion 2006-06 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
to establish whether OK432 sclerotherapy is an effective form of treatment for lymphatic malformations versus the traditional form of treatment, which is surgical excision. | indefinate

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Smith, Study Chair — University of Iowa
Locations (13):
- United States (13):
  - Children's Associated Medical Group, San Diego, California
  - Children's Hospital of Denver, Denver, Colorado
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - All Children's Hospital, St. Petersburg, Florida
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Children's Hospitals and Clinics - Minneapolis, Minneapolis, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Vanderbilt University, Nashville, Tennessee
  - Texas Pediatric Otolaryngology Center, Houston, Texas
  - Children's Hospital of the Kings Daughter, Norfolk, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Smith MC, Zimmerman MB, Burke DK, Bauman NM, Sato Y, Smith RJ; OK-432 Collaborative Study Group. Efficacy and safety of OK-432 immunotherapy of lymphatic malformations. Laryngoscope. 2009 Jan;119(1):107-15. doi: 10.1002/lary.20041. PMID 19117316